CLINICAL TRIAL: NCT00000672
Title: An Efficacy Study of 2',3'-Dideoxyinosine (ddI) (BMY-40900) Administered Orally Twice Daily to Zidovudine Intolerant Patients With AIDS or AIDS-Related Complex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: ACTG 118; 070V1; AI454-007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1994-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
AMENDED: 8/29/90 Inclusion of asymptomatic patients with CD4 counts less than 200 cells/mm3. Standardization of baseline evaluation schedule to allow 14 days prior to study dosing. Reduction in frequency and intensity of follow-up evaluations. Standardization of study endpoints. Inclusion of toxicity scoring and management for amylase and triglyceride elevations. Clarification of concomitant medication use. Original design: To determine the effectiveness of didanosine (ddI) in patients with AIDS or advanced AIDS related complex (ARC) who have documented hematologic intolerance to zidovudine (AZT) therapy. To determine if the efficacy of ddI increases with increasing doses.

AZT is effective in reducing mortality in patients with AIDS who receive the drug after the first episode of Pneumocystis carinii pneumonia (PCP) and in patients with advanced ARC. However, AZT therapy has been associated with significant toxicities. In addition, the effectiveness of AZT appears to decrease during the second and third years of therapy. For these reasons, the development of alternative therapy that would be at least as effective but less toxic is of great importance. The drug ddI is an antiviral agent that inhibits replication (reproduction) of HIV with less apparent toxicity than AZT. The major dose-limiting toxicities found in the Phase I studies have been pains in the feet and legs of 2 patients initially receiving 12 mg/kg/day and 12 patients receiving daily doses of 25.8 to 51.2 mg/kg; symptoms began 8 to 27 weeks after initiating ddI treatment. These neuropathy-like symptoms have generally not been associated with significant abnormalities in nerve conduction studies and patients have reported marked improvement in symptoms within 1 to 2 weeks of discontinuing ddI. Some patients have resumed ddI treatment at a reduced dose after resolution of their symptoms. Studies indicate that ddI remains active in the body for at least 12 hours. This indicates that benefits of ddI might be achieved with a low frequency of drug administration.

DETAILED DESCRIPTION:
AZT is effective in reducing mortality in patients with AIDS who receive the drug after the first episode of Pneumocystis carinii pneumonia (PCP) and in patients with advanced ARC. However, AZT therapy has been associated with significant toxicities. In addition, the effectiveness of AZT appears to decrease during the second and third years of therapy. For these reasons, the development of alternative therapy that would be at least as effective but less toxic is of great importance. The drug ddI is an antiviral agent that inhibits replication (reproduction) of HIV with less apparent toxicity than AZT. The major dose-limiting toxicities found in the Phase I studies have been pains in the feet and legs of 2 patients initially receiving 12 mg/kg/day and 12 patients receiving daily doses of 25.8 to 51.2 mg/kg; symptoms began 8 to 27 weeks after initiating ddI treatment. These neuropathy-like symptoms have generally not been associated with significant abnormalities in nerve conduction studies and patients have reported marked improvement in symptoms within 1 to 2 weeks of discontinuing ddI. Some patients have resumed ddI treatment at a reduced dose after resolution of their symptoms. Studies indicate that ddI remains active in the body for at least 12 hours. This indicates that benefits of ddI might be achieved with a low frequency of drug administration.

Patients are randomized to one of three ddI treatment groups; within each group, doses will be adjusted according to patient's weight at study entry. Stratification is by diagnosis of AIDS or AIDS related complex (ARC) and Medical Center. Data will be tabulated for the Data and Safety Monitoring Board at 3 month intervals.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Aerosolized pentamidine (300 mg every 4 weeks). In the event of physiological intolerance, alternative PCP prophylaxis may be trimethoprim/sulfamethoxazole 1 DS tab per day or dapsone 50 - 100 mg per day.

Allowed:

* Chronic suppressive treatment for toxoplasmosis, Pneumocystis carinii pneumonia (PCP), cryptococcal meningitis, herpes simplex virus, cytomegalovirus, coccidioidomycosis, and histoplasmosis (absorption of ketoconazole or dapsone may be inhibited if given at the same time as the buffered solution of ddI, and should be taken 2 hours before or 2 hours after taking ddI; oral acidifying agents are not allowed). Isoniazid is permitted only if no acceptable alternative therapy is available. Metronidazole may be used for single courses not to exceed 14 days within consecutive 90 day intervals, the first of which begins at the initiation of the study. Erythropoietin for patients under the relevant treatment IND. Intravenous acyclovir for short courses of therapy.

Patients must:

* Have documented hematologic intolerance to zidovudine (AZT).
* Have the diagnosis of AIDS or advanced AIDS related complex (ARC).
* Have ended treatment for acute Pneumocystis carinii pneumonia (PCP) at least 2 weeks before study entry.

Have previous intolerance on at least two courses of AZT therapy (one of which must have been at daily doses of 500 mg of AZT or less).

* Be able to provide informed consent (and/or guardian as appropriate).
* Be available for follow-up for at least 6 months.
* Have baseline laboratory values as measured within 7 days before initial drug dosing.
* Allowed:
* Development of new opportunistic infections during the study - patients remain in the protocol.

Prior Medication:

Required:

* Prior use and intolerance to zidovudine (AZT).
* Allowed:
* Intralesional agents.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Presence of Kaposi's sarcoma (KS) with known or suspected visceral disease or where KS requires chemotherapy.
* Active AIDS defining opportunistic infections not specifically allowed.
* Intractable diarrhea.
* Stage 2 AIDS-dementia complex.
* History of intolerance to aerosolized pentamidine.
* Grade 2 neuropathy, based on the Neuropathy Targeted Symptom Questionnaire, or any moderate abnormality indicative of peripheral neuropathy, particularly impaired sensation of sharp pain, light touch, or vibration in the lower extremities, distal extremity weakness, or distal extremity hyporeflexia.
* Prior history of acute or chronic pancreatitis.
* History of seizures within past 2 years or currently requiring anticonvulsants for control.
* Any other clinical conditions or prior therapy which, in the opinion of the investigator, would make the patient unsuitable for study or unable to comply with the dosing requirements.

Concurrent Medication:

Excluded:

* Isoniazid (INH).

Patients with the following are excluded:

* Active AIDS-defining opportunistic infections not specifically allowed.
* Intractable diarrhea.
* AIDS-dementia complex = or > stage 2.
* History of intolerance to aerosolized pentamidine. Grade 2 neuropathy, based on the Neuropathy Targeted Symptom Questionnaire, or any moderate abnormality indicative of peripheral neuropathy, particularly impaired sensation of sharp pain, light touch, or vibration in the lower extremities, distal extremity weakness, or distal extremity hyporeflexia.
* Prior history of acute or chronic pancreatitis.
* History of seizures within past 2 years or currently requiring anticonvulsants for control.
* Any other clinical conditions or prior therapy which, in the opinion of the investigator, would make the patient unsuitable for study or unable to comply with the dosing requirements.
* Previous participation in any Phase I ddI study.
* Life expectancy < 6 months.

Prior Medication:

Excluded:

* Chronic therapy for cytomegalovirus infection with ganciclovir.
* ddI.
* d4T.
* ddC.

Excluded within 2 weeks of study entry:

* Zidovudine (AZT).

Excluded within 1 month of study entry:

* Therapy with any other antiretroviral drug or investigational agent not specifically allowed, including interferon and immunomodulating drugs.
* Ganciclovir.
* Neurotoxic drugs.

Excluded within 3 months of study entry:

* Ribavirin.
* Cytotoxic anticancer therapy.

Prior Treatment:

Excluded within 2 weeks of study randomization:

* Transfusion.

Active alcohol or drug abuse that is sufficient, in investigator's opinion, to prevent adequate compliance with study therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660
Dates: Primary Completion 1993-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JD Allan, Study Chair; J Groopman, Study Chair; M Seidlin, Study Chair
Locations (67):
- United States (66):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford Univ School of Medicine, Stanford, California
  - Olive View Med Ctr, Sylmar, California
  - Sepulveda Veterans Adm Med Ctr / Olive View Med Ctr, Sylmar, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Mountain States Regional Hemophilia Ctr / Univ of Colorado, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - G E Morey Jr, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of South Florida, Tampa, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Edward Hines Veterans Administration Hosp, Hines, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Louisiana Comprehensive Hemophilia Care Ctr, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Med Ctr of Central Massachusetts, Worcester, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Nebraska Regional Hemophilia Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Hemophilia Ctr / Mount Sinai Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Bowman Gray School of Medicine / Wake Forest Univ, Winston-Salem, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Univ of Washington, Seattle, Washington
  - Great Lakes Hemophilia Foundation, Milwaukee, Wisconsin
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Fichtenbaum CJ, Clifford DB, Powderly WG. Risk factors for dideoxynucleoside-induced toxic neuropathy in patients with the human immunodeficiency virus infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Oct 1;10(2):169-74. doi: 10.1097/00042560-199510020-00009. PMID 7552481
- [Background] Kozal MJ, Kroodsma K, Winters MA, Shafer RW, Efron B, Katzenstein DA, Merigan TC. Didanosine resistance in HIV-infected patients switched from zidovudine to didanosine monotherapy. Ann Intern Med. 1994 Aug 15;121(4):263-8. doi: 10.7326/0003-4819-121-4-199408150-00005. PMID 7518658
- [Background] Reddy MM, Winger EE, Hargrove D, McHugh T, McKinley GF, Grieco MH. An improved method for monitoring efficacy of anti-retroviral therapy in HIV-infected individuals: a highly sensitive HIV p24 antigen assay. J Clin Lab Anal. 1992;6(3):125-9. doi: 10.1002/jcla.1860060305. PMID 1506978
- [Background] Grieco MH, McKinley GF, Reddy MM. Effect of 2',3',-dideoxyinosine on HIV P24 antigen, beta2-microglobulin, neopterin,SCD8,SCD4,and SIL2R levels in patients with ARC or AIDS. Int Conf AIDS. 1991 Jun 16-21;7(2):199 (abstract no WB2069)
- [Background] Bozzette SA, Hays RD, Berry SH, Kanouse DE. A Perceived Health Index for use in persons with advanced HIV disease: derivation, reliability, and validity. Med Care. 1994 Jul;32(7):716-31. doi: 10.1097/00005650-199407000-00005. PMID 8028406
- [Background] Fiscus SA, Heggem-Snow A, Troiani L, Wallmark E, Folds JD, Sheff B, van der Horst CM. Transient high titers of HIV-1 in plasma and progression of disease. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 May 1;9(1):51-7. PMID 7712235
- [Background] Spino C, Kahn JO, Dolin R, Phair JP. Predictors of survival in HIV-infected persons with 50 or fewer CD4 cells/mm3. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Aug 15;15(5):346-55. doi: 10.1097/00042560-199708150-00004. PMID 9342254
- [Background] Allan JD, DeGruttola V, Cross A, McLaren C, Seidlin M, Pettinelli C. An efficacy study of 2'3'-dideoxyinosine [ddI](BMY-40900) administered orally twice daily to zidovudine intolerant patients with HIV infection (ACTG 118). The AIDS Clinical Trials Group. Int Conf AIDS. 1993 Jun 6-11;9(1):67 (abstract no WS-B24-2)
- [Background] Sharma PL, Chatis PA, Dogon AL, Mayers DL, McCutchan FE, Page C, Crumpacker CS. AZT-related mutation Lys70Arg in reverse transcriptase of human immunodeficiency virus type 1 confers decrease in susceptibility to ddATP in in vitro RT inhibition assay. Virology. 1996 Sep 15;223(2):365-9. doi: 10.1006/viro.1996.0488. PMID 8806572